CLINICAL TRIAL: NCT05759390
Title: Role of Ultrasound Elastography in Differentiation of Peripheral Lung Lesions
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Waleed Gamal Elddin Khaleel, Lecturer of chest diseases and tuberculosis, Assiut University
Other Study IDs: Elastography in Lung
Record Dates: First submitted 2023-02-26; First posted 2023-03-08 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Lung Diseases
Keywords: Ultrasound elastography; lung lesions
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasound elastography — Using an ultrasound scanner for chest ultrasound examinations. If patients has multiple sub pleural lung lesions, the largest and most approachable lesion to perform 2 Dimensions- shear wave elastography (2D-SWE) will be chosen.

SUMMARY:
Advancements in imaging capacities and the development of a precise puncture-guiding transducer have made transthoracic ultrasonography a useful diagnostic tool for evaluating peripheral subpleural lung tumours. Different human tissues have varying levels of elasticity because of the properties of the extracellular matrix.

Pleural two-dimensional (2D) shear-wave elastography (SWE) can be used to differentiate between malignant pleural effusion and benign pleural disease.

Transthoracic 2D-SWE uses acoustic radiation force and assesses the velocity of tissue displacement propagation in multiple focal zones. The shear waves are monitored in 2D by creating a near-cylindrical shear-wave cone, enabling measurement of the shear-wave speed or Young's modulus (E) on a colour quantitative elastogram. Based on the hypothesis that transthoracic 2D-SWE could add accurate tissue stiffness information to B-mode grayscale ultrasound images and help in differentiating lung malignancy from benign lung lesions.

DETAILED DESCRIPTION:
B-mode grayscale images will be used by ultrasound to assess peripheral lung lesions. Information including size, location, and intercostal chest wall thickness will be collected. Then, Investigators will use transthoracic 2D-SWE to assess those lesions.

Investigators intend to use regions of interest (ROIs) with 3-mm diameter, and select up to four ROIs with the highest mean elasticity values. the average as the final value will be calculated. If patients had multiple sub-pleural lung lesions, the largest and the most approachable one will be chosen to perform 2D-SWE. Final diagnosis will be made via appropriate diagnostic modalities including computed tomography of chest, microbiological results and guided biopsies if indicated.

ELIGIBILITY:
Inclusion Criteria:

* Radiographic evidence of pulmonary lesions

Exclusion Criteria:

* Patients less than 18 years.
* Patients refusing to participate in the study.
* Inability to hold breath for at least 5 s.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients aged more than 18, presented with peripheral lung lesions not readily diagnosed.
  ultrasound elastography used to differentiate benign from malignant lung lesions
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Evaluate the predictive value of transthoracic 2 Dimension- Shear Wave Elastography (2D-SWE) in the diagnosis of peripheral lung lesions. | 1 MONTH
  Peripheral lung lesions evaluated using 2 Dimension- Shear Wave Elastography to differentiate between benign and malignant lung lesions comparing the results to definitive diagnostic method either microbiological results and pathological specimens obtained by biopsy if indicated.

CONTACTS AND LOCATIONS:
Overall Officials: Waleed Gamal Elddin, Lecturer, Principal Investigator — Assiut university, Egypt
Locations (1):
- Assiut university hospitals, Asyut, Egypt

REFERENCES:
- [Background] Jiang B, Li XL, Yin Y, Zhang Q, Zang T, Song WS, Wang XM, Kang J, Herth FJF, Hou G. Ultrasound elastography: a novel tool for the differential diagnosis of pleural effusion. Eur Respir J. 2019 Aug 22;54(2):1802018. doi: 10.1183/13993003.02018-2018. Print 2019 Aug. PMID 31151959
- [Background] Bedawi EO, Guinde J, Rahman NM, Astoul P. Advances in pleural infection and malignancy. Eur Respir Rev. 2021 Jan 13;30(159):200002. doi: 10.1183/16000617.0002-2020. Print 2021 Mar 31. PMID 33650525